CLINICAL TRIAL: NCT02272595
Title: A Study to Select Rational Therapeutics Based on the Analysis of Matched Tumor and Normal Biopsies in Subjects With Advanced Malignancies
Brief Title: Rational Therapeutics Based on Matched Tumor and Normal Tissue
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: PA12-0381
Record Dates: First submitted 2014-10-20; First posted 2014-10-23 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancers
Keywords: Biologic Markers; Molecular testing; Advanced cancers; Molecular information; Molecular profiling; Genetic Mutation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (about 2 teaspoons) drawn initially and again about 2-3 weeks after chosen treatment begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A - Treatment Based on Genetic Mutation: Participant's molecular profile shows that they have a gene mutation that may benefit from study drugs that are believed to target their gene mutation. Participant assigned to Arm A and will receive these targeted drugs.
  Interventions: Other: Treatment Based on Genetic Mutation
- Arm B - Treatment Based on No Genetic Mutation: Participant's molecular profile shows that they do not have a gene mutation. Participant assigned to Arm B in which doctor chooses a therapy based on other studies rather than gene mutation.
  Interventions: Other: Treatment Based on No Genetic Mutation

INTERVENTIONS:
Other: Treatment Based on Genetic Mutation — Participant's molecular profile shows that they have a gene mutation that may benefit from study drugs that are believed to target their gene mutation. Participant assigned to Arm A and will receive these targeted drugs.
  Groups: Arm A - Treatment Based on Genetic Mutation
Other: Treatment Based on No Genetic Mutation — Participant's molecular profile shows that they do not have a gene mutation. Participant assigned to Arm B in which doctor chooses a therapy based on other studies rather than gene mutation.
  Groups: Arm B - Treatment Based on No Genetic Mutation

SUMMARY:
The goal of this laboratory research study is to learn if using molecular information (matched therapy) or not using molecular information and having the study doctor choose the therapy based on your past experience are more effective ways to choose the best cancer treatment for you.

This is an investigational study.

Up to 200 participants will take part in this study. Up to 50 will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
If you agree to take part in this study, your tumor tissue and blood samples will be tested for molecular profiling. Molecular profiling is the classification of tissue based on the expression of certain genes within a tumor compared to normal tissue. This may be used to predict how the tumor responds to therapy. Your doctor may use the results of the molecular profiling to help decide which treatment might be the most beneficial for the disease.

Study Procedures:

Blood (about 2 teaspoons) will be drawn and you will have a tumor biopsy and a biopsy of normal tissue when you enroll in this study. Blood (about 2 teaspoons) will be drawn again about 2-3 weeks after you begin treatment. The type of biopsy you have will depend on the type of disease you have. The risks of this procedure will be discussed in more detail with you.

If there is not enough tissue with which the study doctor can perform the study tests (described below), you may need to have a second biopsy. The study staff will discuss this with you if it is needed.

Treatment Arms:

A series of tests to find which gene mutations you have, if any, will be performed. Depending on the results of your molecular testing, you may be enrolled on 1 of 2 arms.

If your molecular profile shows that you have a gene mutation that may benefit from study drugs that are believed to target your gene mutation, you will be enrolled in Arm A and will receive these targeted drugs.

If your molecular profile shows that you do not have a gene mutation, you will be enrolled in Arm B. In Arm B, the doctor will choose a therapy based on other studies rather than gene mutation.

Length of Study:

This study will last about 2 years. Your participation on this study will be complete after the last blood draw and tumor biopsy is collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Any histologic type of metastatic cancer, (except for lung and brain at US sites), in which histologic normal counterpart can be obtained. See list of cancer types included in the trial in Appendix 1.
3. Progression by RECIST (Response Evaluation Criteria In Solid Tumors) or other criteria on at least one prior regimen for advanced disease
4. Ability to undergo a biopsy or surgical procedure to obtain fresh tumor biopsy paired with its normal counterpart
5. Age from 18 years
6. Life expectancy of at least 3 months
7. ECOG Performance status of 0 to 1
8. Measurable or evaluable disease according to RECIST 1.1 criteria
9. For US sites only: advanced cancer patients that have exhausted all effective therapy for their disease and have progressed after previous line of therapy (documented disease progression under last treatment received) and conventional methods of assigning new therapy would not be expected to increase survival by more than 3 months.

Exclusion Criteria:

1. For US sites only: Any patient that might require a lung or brain biopsy are excluded
2. Alteration of organ function or hematopoietic function as defined by the following criteria:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) >2.5 x upper limit of normal (ULN), except for patients with liver metastases, for which AST and ALT > 5.0 ULN is the exclusion criteria.
   2. Bilirubin > 2.0 ULN to allow for Gilberts
   3. Polynuclear neutrophil < 1.5 x 109/L
   4. Platelets < 100 x 10 9/L
   5. Hemoglobin < 90 g/L
   6. Creatinine > 1.5 ULN

   i. Calcemia > 1.5 ULN g. Phosphatemia > 1.5 ULN
3. Coagulation abnormality prohibiting a biopsy
4. Symptomatic or progressive brain metastases detected by radio imaging, or meningeal
5. Patient who received a personalized therapeutic treatment based on molecular anomaly during the treatment period immediately prior to the WINTHER directed treatment (defining the PFS1). Hormonal therapy may be continued during WINTHER suggested therapy. The exclusion of prior matched targeted therapy includes but is not limited to all targeted therapeutics that are EMA approved and genomically matched to patients. If there are questions about whether or not a prior therapy is a matched targeted treatment it will be agreed on by discussion between PIs who are also Clinical Management Committee members; the resolution should take place prior to starting Winther directed treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients from University of Texas MD Anderson Cancer Center in Houston, Texas, Cancer Institute Gustave Roussy in Villejuif, France, Vall D'Hebron University Hospital in Barcelona, Spain, and Chaim Sheba Medical Center at Tel Hasomer in Ramat Gan, Israel
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 - 3 weeks after treatment begins
  Progression-free survival (PFS) of the last therapeutic line (PFS1) before entering into study, with the PFS2 under study treatment. A clinical meaningful improvement is defined as demonstrating a PFS ratio (PFS2/PFS1) of being 1.5 or better.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Cancer Institute Gustave Roussy, Villejuif, France
- Chaim Sheba Medical Center at Tel Hasomer, Ramat Gan, Israel
- Vall D'Hebron University Hospital, Barcelona, Spain

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org